CLINICAL TRIAL: NCT00499447
Title: A Phase II Study of Radiofrequency Ablation Combined With External Beam Radiation Therapy for Patients With Medically Inoperable Non-Small Cell Lung Cancer (Stage Ia and Select Ib) and the Predictive Value of Positron Emission Tomography
Brief Title: Radiofrequency Ablation and External-Beam Radiation Therapy in Treating Patients With Stage I Non-Small Cell Lung Cancer That Cannot Be Removed by Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000555009; CCCWFU 62306 (Other: CCCWFU); IRB00001334 (Other: WFUHS IRB)
Record Dates: First submitted 2007-07-10; First posted 2007-07-11 (Estimated); Results first posted 2013-03-01 (Estimated); Last update posted 2019-05-08 (Actual); Status verified 2016-03

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; adenocarcinoma of the lung; adenosquamous cell lung cancer; large cell lung cancer; squamous cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — Radiofrequency Ablation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Radiofrequency Ablation with External Beam Radiation (Experimental): Radiofrequency Ablation (RFA)under computerized tomography guidance followed 3-4 weeks later with External Beam Radiation Therapy
  Interventions: Procedure: radiofrequency ablation; Radiation: radiation therapy

INTERVENTIONS:
Procedure: radiofrequency ablation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiofrequency ablation uses a high-frequency electric current to kill tumor cells. External-beam radiation therapy uses high-energy x-rays to kill tumor cells. Giving radiofrequency ablation together with radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving radiofrequency ablation together with external-beam radiation therapy works in treating patients with stage I non-small cell lung cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine progession free survivial rates in patients with inoperable stage IA and select stage IB non-small cell lung cancer treated with external-beam radiation therapy and radiofrequency ablation (RFA).

Secondary

* To determine the acute and late toxicity of combining RFA with external-beam radiation therapy.
* To determine the patterns of failure at time of first relapse.
* To determine the rate of overall survival at 1 and 2 years after treatment.
* To evaluate the ability of peak standard uptake value (SUV) and max SUV obtained prior to RFA to predict local control and time to progression.
* To measure post RFA/simulation (treatment planning) PET max and peak SUV's and correlate this data with local control at 1 and 2 years.
* To evaluate the ability of peak and max SUV's for fludeoxyglucose F 18 obtained shortly after radiotherapy (post-treatment) to predict local control and time to progression.
* To evaluate PET-CT data and its utility in guiding radiation therapy treatment planning.
* To explore the use of dual time point imaging PET data obtained to predict local control and also to differentiate between recurrence versus inflammation when applicable.
* To assess physical function as a prognostic measure, and to determine the impact of treatment on physical function.
* To evaluate the impact of treatment on generic and disease-specific quality of life.

OUTLINE: Patients undergo fludeoxyglucose F18 positron emission tomography (FDG-PET) and CT scan at baseline. Patients then undergo radiofrequency ablation (RFA). Beginning within 5 weeks after completion of RFA, patients undergo external-beam radiation therapy once daily, 5 days a week, for 5-6 weeks. FDG-PET/CT scan is repeated 3-4 weeks after RFA and 12-16 weeks after completion of external-beam radiation therapy.

Quality of life is assessed at baseline, during treatment, and at 16 weeks and at 1 year after completion of treatment.

After completion of study treatment, patients are followed periodically for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-small cell lung cancer

  * Cytology or biopsy-proven disease
  * Stage IA (T1N0M0) or select stage IB (T2N0M0 because of visceral pleural involvement or size ≥ 3.0 cm)
  * Tumor size ≤ 3.5 cm
* No bronchioloalveolar carcinoma
* Node-negative patients will have hilar or mediastinal lymph nodes ≤ 1.5 cm and no clinically suspicious uptake on fludeoxyglucose F 18 (FDG)-PET in those areas

  * Patients with > 1.5 cm lymph nodes and clinically suspicious FDG-PET uptake will still be eligible if directed tissue biopsy or needle aspiration of abnormally identified area are negative for cancer
  * Patients with > 1.5 cm and < 2.0 cm lymph nodes and no clinically suspicious FDG-PET uptake in those areas will still be eligible
* All patients are required to have been evaluated by a thoracic surgeon and have either refused surgery or been deemed medically inoperable due to comorbid conditions
* CT images of the chest must be reviewed by an experienced interventional radiologist and the target lesion must be determined to be in a location where radiofrequency ablation is technically achievable based on the proximity of adjacent organs and structures
* Any patient with suspected M1 disease based on pre-treatment PET-CT imaging should have biopsy if possible

  * If the biopsy is positive, the patient should be treated as per the clinician's preference off of this protocol
  * If the biopsy is negative and representative of the lesion in question then the patient may be treated as per this protocol
  * If the biopsy is non-diagnostic, consideration should be given to repeat biopsy
  * If the repeat biopsy remains non-diagnostic or a biopsy is not feasible than the patient will not be eligible for this protocol and should be treated per the clinician's preference

PATIENT CHARACTERISTICS:

* Inclusion Criteria:

  * ECOG performance status 0-2
  * Women of childbearing potential must have a negative pregnancy test
  * Fertile women must use effective contraception
* Exclusion Criteria:

  * History of prior malignancy within the past 2 years except for curatively treated basal cell carcinoma of the skin, cervical intra-epithelial neoplasia, T1N0 squamous cell carcinoma of the larynx, or localized prostate cancer with a current PSA level < 1.0 mg/dL on 2 successive evaluations, at least 3 months apart, with the most recent evaluation no more than 4 weeks prior to study entry
  * Pregnant or lactating women

PRIOR CONCURRENT THERAPY:

* Exclusion Criteria:

  * Previous chest radiation to the lung or mediastinum
  * Patients must not receive other concurrent anticancer therapies while on protocol including any of the following:

    * Radiotherapy
    * Radiofrequency ablation
    * Other antineoplastic interventional radiology techniques
    * Chemotherapy
    * Biological therapy
    * Vaccine therapy
    * Surgery

      * Surgical treatment of nonmelanomatous skin cancer or ≤ T1 urothelial cell carcinoma allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-05 (Actual); Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Blackstock, MD, Study Chair — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Radiation Oncology Clinic at the Comprehensive Cancer Center of Wake Forest University.
Period: Overall Study
Arm/Group | Radiofrequency Ablation Combined With External
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Radiofrequency Ablation Combined With External
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.5 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Two Year Progression Free Survival Rate
Description: the number of patients surviving progression-free at two years.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Radiofrequency Ablation Combined With External
Number analyzed (Participants) | 13
participants | 8

ADVERSE EVENTS:
Arm/Group | Radiofrequency Ablation Combined With External
Serious Adverse Events (participants affected / at risk) | 8/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiofrequency Ablation Combined With External (N=12)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Carbon monoxide diffusion (Investigations) | 4 (4)
hyperglycemia (Investigations) | 2 (2)
decreased forced expiratory volume (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Lymphopenia (Investigations) | 4 (4)
Lung infection (Infections and infestations) | 1 (1)
Burn (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiofrequency Ablation Combined With External (N=12)
Low WBC (Investigations) | 3 (3)
low Platelets (Investigations) | 3 (3)
Low Hemoglobin (Investigations) | 8 (11)
Hemorrhage/Bleeding - Other (Vascular disorders) | 2 (2)
Anorexia (General disorders) | 1 (1)
Alkaline phosphatase (Investigations) | 1 (1)
Urinary retention (including neurogenic bladder) (General disorders) | 1 (1)
Dyspnea (Reproductive system and breast disorders) | 4 (5)
Carbon monoxide diffusion (Investigations) | 8 (8)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hypertension (General disorders) | 2 (2)
Neuropathy: motor (Nervous system disorders) | 1 (1)
Low ANC (Investigations) | 1 (1)
Insomnia (General disorders) | 1 (1)
Rigors/chills (General disorders) | 1 (1)
Sweating (General disorders) | 1 (1)
Fatigue (General disorders) | 5 (6)
hyperglycemia (Investigations) | 8 (10)
hypoglycemia (Investigations) | 2 (2)
hypocalcemia (Investigations) | 2 (2)
hypomagnesemia (Investigations) | 1 (1)
hyponatremia (Investigations) | 1 (1)
hypokalemia (Investigations) | 2 (2)
hypoalbuminemia (Investigations) | 4 (4)
hyperbilirubinemia (Investigations) | 1 (1)
serum glutamic oxaloacetic transaminase (Investigations) | 1 (1)
hypernatremia (Investigations) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1)
Ocular/Visual - Other (Eye disorders) | 1 (1)
Dysphagia (General disorders) | 2 (2)
Fever without neutropenia (General disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Edema: limb (Vascular disorders) | 1 (1)
Heartburn/dyspepsia (General disorders) | 1 (1)
Hypoxia (Investigations) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Partial Thromboplastin Time (Investigations) | 1 (1)
Ataxia (General disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pain: Back (General disorders) | 2 (2)
Amylase (Investigations) | 1 (1)
"Fistula, pulmonary/upper respiratory: Bronchus" (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchospasm wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain: Chest/thorax (General disorders) | 2 (2)
Pain: Chest wall (General disorders) | 5 (7)
decreased forced expiratory volume (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
hypertriglyceridemia (Investigations) | 1 (1)
Injection site reaction (Immune system disorders) | 1 (1)
Lymphopenia (Investigations) | 2 (2)
Memory impairment (General disorders) | 1 (1)
Pain: Muscle (General disorders) | 1 (1)
Nail changes (General disorders) | 1 (1)
Ulcer Esophagus (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Esophagitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Hemorrhage Lung (Vascular disorders) | 2 (2)
Soft tissue necrosis Thorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vital capacity (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Infection with unknown ANC Lung (pneumonia) (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
adverse events were tracked in two cycles, one during treatment and one longer term

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes